CLINICAL TRIAL: NCT00028951
Title: A Phase III Clinical Trial Use of TISSEEL VH Fibrin Sealant to Reduce Lymphedema Incidence After Inguinal Lymph Node Dissection Performed in the Management of Vulvar Malignancies
Brief Title: Fibrin Sealant in Decreasing Lymphedema Following Surgery to Remove Lymph Nodes in Patients With Cancer of the Vulva
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000069149; GOG-0195; NCI-P01-0201
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2005-12

CONDITIONS: Lymphedema; Perioperative/Postoperative Complications; Vulvar Cancer
Keywords: lymphedema; perioperative/postoperative complications; stage I vulvar cancer; stage II vulvar cancer; stage III vulvar cancer; stage IVB vulvar cancer
MeSH Terms: conditions — Lymphedema; Postoperative Complications; Vulvar Neoplasms | interventions — Fibrin Tissue Adhesive; Wound Closure Techniques

INTERVENTIONS:
Drug: fibrin sealant
Procedure: surgical wound closure

SUMMARY:
RATIONALE: Fibrin sealant may decrease lymphedema following surgery to remove lymph nodes in the groin by helping to seal the lymphatic vessels. It is not yet known if fibrin sealant is effective in decreasing lymphedema following surgery to remove lymph nodes.

PURPOSE: Randomized phase III trial to determine the effectiveness of fibrin sealant in reducing lymphedema following surgical removal of lymph nodes in patients who have cancer of the vulva.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of lymphedema of the lower extremity after lymph node dissection in patients with vulvar malignancies treated with fibrin sealant vs standard care.
* Compare the frequency of surgical complications in patients treated with fibrin sealant vs standard care.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: After radical vulvectomy or hemivulvectomy and lymphadenectomy, patients receive fibrin sealant to surgical site.
* Arm II: After surgery, patients receive standard care for closure of surgical site.

Lymphedema is assessed at time of drain removal, at week 6, and then at months 3 and 6.

Patients are followed at week 6 and at months 3 and 6.

PROJECTED ACCRUAL: A total of 120-130 patients (60-65 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of vulvar malignancy

  * Stage I-IVB
* Planned radical vulvectomy or hemivulvectomy AND
* Ipsilateral or bilateral inguinal lymphadenectomy
* Presence of groin node metastases is allowed
* No primary or secondary lymphedema of the lower extremities

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* GOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* No bleeding disorder

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Albumin at least 3.0 g/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No prior lower extremity deep vein thrombosis

Other:

* No known sensitivity or anaphylaxis to bovine-derived products
* No known prior exposure to fibrin tissue adhesive
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No nonhealing ulcer or chronic infection of the lower extremity, including superficial phlebitis
* No prior fracture of any portion of either leg
* Preoperative circumferential measurements of legs must differ by less than 3 cm
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for a prior malignancy
* Concurrent adjuvant chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for a prior malignancy
* No prior radiotherapy to pelvis, abdomen, inguinal area, or lower extremity

Surgery:

* See Disease Characteristics
* No prior inguinal surgery
* No prior surgery to veins or arteries of either leg
* No other concurrent elective surgery during same operative event as inguinal lymphadenectomy

Other:

* At least 30 days since prior investigational products or devices
* At least 7 days since prior anticoagulants
* Concurrent enrollment on GOG-0173 or other adjuvant treatment protocols is allowed
* No other concurrent investigational products or devices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Incidence of lymphedema of the lower extremity at 1 week, 6 weeks, 3 months, and 6 months postoperatively

SECONDARY OUTCOMES:
Frequency of surgical complications at 1 week, 6 weeks, 3 months, and 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jay W. Carlson, DO, Study Chair — Gynecologic Oncology of West Michigan
Locations (49):
- United States (49):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - Medical Center Hospital of Vermont Campus, Burlington, Vermont
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Result] Carlson JW, Kauderer J, Walker JL, Gold MA, O'Malley D, Tuller E, Clarke-Pearson DL; Gynecologic Oncology Group. A randomized phase III trial of VH fibrin sealant to reduce lymphedema after inguinal lymph node dissection: a Gynecologic Oncology Group study. Gynecol Oncol. 2008 Jul;110(1):76-82. doi: 10.1016/j.ygyno.2008.03.005. Epub 2008 May 15. PMID 18482765
- [Result] Carlson J, Kauderer J, Walker J, et al.: Phase III trial of Tisseel to reduce lymphedema after inguinal lymph node dissection: a Gynecologic Oncology Group study. [Abstract] Society of Gynecologic Oncologists, 2007 Annual Meeting on Women's Cancer, March 3-7, 2007, San Diego, CA. A-228, 2007.